CLINICAL TRIAL: NCT07379268
Title: Study Protocol for Evaluating the Efficacy of Anti-HER-2 Antibody-Drug Conjugates (ADC) in Locally Advanced or Metastatic Bladder Cancer Based on Organoid Technology.
Brief Title: Evaluation of the Efficacy of Anti-HER2 Antibody-Drug Conjugates (ADC) in Locally Advanced or Metastatic Bladder Cancer Based on Organoid Technology.
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: The Second Hospital of Shandong University (Other); Qianfoshan Hospital (Other); Shandong Provincial Hospital (Other Government); Shandong Province Third hospital (Other); Taian City Central Hospital (Other); Weifang People's Hospital (Other); Binzhou Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Jining First People's Hospital (Other); Liaocheng People's Hospital (Other); Linyi People's Hospital (Other); Yantai Yuhuangding Hospital (Other); Zibo Central Hospital (Other Government); Dezhou Hospital Qilu Hospital of Shandong University (Other); Zaozhuang Municipal Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202411-010-1
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
Keywords: Organoid; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Using tumor organoid drug sensitivity tests to detect the sensitivity of patients' tumor cells to the anti-HER2-ADC drug vedicitumumab, the anti-HER2-ADC treatment regimen is only used for patients whose sensitivity to the drug has been confirmed through tumor organoid drug sensitivity testing.
  Interventions: Other: Organoid culture
- Control group: Select bladder cancer patients diagnosed during the same period who received anti-HER2-ADC drugs based on HER2 protein overexpression (immunohistochemistry IHC 2 and 3) as the control group.

INTERVENTIONS:
Other: Organoid culture — Organoid culture of tumor tissue obtained during patient surgery
  Groups: Experimental group

SUMMARY:
This study, through a clinical controlled trial, compares the one-year, two-year, and three-year overall survival rates of patients in the treatment group guided by organoid drug sensitivity intervention with those of patients whose medication was based on HER-2 protein expression levels (IHC method). Univariate Kaplan-Meier survival analysis was used to compare differences in overall survival between the two groups. The study aims to evaluate the application value of tumor organoid drug sensitivity testing in guiding anti-HER2-ADC drug treatment for bladder cancer.

DETAILED DESCRIPTION:
1. Research Background (Rationale and Significance Based on Domestic and International Research Status)

   Bladder cancer is a malignant tumor originating from the bladder urothelium and ranks first in incidence among urogenital tumors in China. Urothelial carcinoma is the most common type, accounting for over 90% of bladder cancer cases [1]. Approximately 5% of bladder cancer patients are diagnosed with metastatic disease, termed metastatic bladder cancer (MBC) [2-4]. Studies have shown that the median progression-free survival (PFS) for MBC patients is 7 months, and the median overall survival (OS) is 15 months [5, 6].

   For patients with unresectable locally advanced or distant metastatic bladder cancer, platinum-based combination chemotherapy (CC) remains the standard first-line treatment [7]. In recent years, with continuous advancements in medical technology, the emergence of novel chemotherapeutic agents, targeted drugs, and immune checkpoint inhibitors has significantly increased the therapeutic options available after progression on first-line chemotherapy for MBC, yielding promising efficacy [8]. Anti-HER2 antibody-drug conjugates (ADCs), represented by trastuzumab-based therapies, are among these options. Human epidermal growth factor receptor 2 (HER2) is a transmembrane tyrosine kinase receptor involved in stimulating cell proliferation, differentiation, and survival [9]. HER2 overexpression plays a significant role in the development and progression of various malignancies, including breast cancer, gastric cancer, and urothelial carcinoma [10], and is often associated with a biologically aggressive tumor phenotype, poor prognosis, increased risk of disease recurrence, and limited benefit from chemotherapy [9, 11-13]. In bladder urothelial carcinoma, the proportion of HER2 protein overexpression (Immunohistochemistry [IHC] 2+ and 3+) ranges from 18.1% to 36% [14-16], and HER2 gene amplification is observed in 10% to 23% of cases [14, 16-17]. Research indicates that anti-HER2 ADC drugs demonstrate good efficacy and safety in treating patients with locally advanced unresectable or metastatic urothelial carcinoma, providing significant clinical benefit for this population [18]. In June 2021, Disitamab Vedotin (RC-48, RemeGen Co., Ltd.) was approved in China for the treatment of HER2-positive locally advanced or metastatic urothelial carcinoma [10]. HER2 protein expression status is typically assessed using IHC [10]. However, there is currently no internationally standardized detection protocol or interpretation criteria for HER2 protein expression status in urothelial carcinoma. This leads to considerable discrepancies in HER2 expression assessment across different clinical centers, directly affecting the selection of patients eligible for anti-HER2 ADC therapy and the standardization of clinical research. Additionally, fluorescence in situ hybridization (FISH) testing for HER2 gene amplification status also holds clinical significance for treatment guidance [10]. Clinical studies suggest that HER2 ADC drugs remain effective in urothelial carcinoma patients with HER2 protein overexpression (IHC 2+) but negative FISH results [18, 19], and clinically, there are patients who benefit despite negative protein detection but positive FISH. These findings indicate that neither IHC nor FISH results alone can fully guide the use of Disitamab Vedotin. When clinical assessment determines a patient's insensitivity to the administered drug, severe toxic side effects have often already occurred, and disease progression may deprive the patient of opportunities for alternative treatments. Therefore, evaluating the response of locally advanced or metastatic bladder cancer patients to anti-HER2 antibody-drug conjugates to guide treatment selection for patients with high drug sensitivity, thereby achieving precise and individualized tumor therapy, has increasingly become a current research focus.

   The realization of precise cancer treatment heavily relies on drug sensitivity testing. Through precise and individualized drug screening experiments, the most effective and least toxic treatment regimen can be identified for each patient before therapy begins. Developing patient-specific treatment plans represents a new research direction for achieving precision treatment in bladder cancer and improving drug efficacy. Previously, commonly used preclinical models included traditional tumor cell lines and patient-derived xenograft (PDX) models. Tumor cell line culture is simple but insufficient to simulate the growth state of tumor cells within the patient's body, and drugs screened using these systems have low clinical translation value. While PDX models can simulate in vivo tumor characteristics and preserve the tumor microenvironment, they have significant limitations, such as relatively low stable engraftment rates, long modeling and evaluation cycles (six months to one year), being time-consuming and labor-intensive, making them difficult to generate and utilize for high-throughput drug screening [20-23]. Therefore, to develop more personalized treatment and prevention strategies tailored to an individual's unique genetic, environmental, and lifestyle characteristics, minimizing risks and optimizing medical intervention outcomes, it is imperative to develop drug sensitivity testing models that can simulate the heterogeneity and complexity of bladder cancer.

   Organoids, specifically Patient-Derived Organoids (PDOs), are three-dimensional organotypic structures formed through the self-assembly of stem cells in vitro. They can differentiate into multiple organ-specific cell types and exhibit cell-cell interactions, cell-extracellular matrix interactions, and spatial organization, thereby recapitulating key functions and structures of real human organs in vitro while maintaining stable phenotypic and genetic characteristics. Compared to two-dimensional tumor cell lines and PDX models, tumor organoids can be cultured directly from a patient's own tissue. These organoids can effectively replicate key properties of the primary tumor, preserve the pathological morphology and biological mechanisms of the patient's tissue, retain tumor heterogeneity and a more authentic tumor microenvironment, and have the advantage of a short growth cycle [24]. This facilitates their use for sensitivity testing of chemotherapy drugs, molecularly targeted agents, and anti-tumor antibodies in clinical cancer patients, predicting patient response to drugs, and holds potential for assisting clinical treatment decision-making.

   In 2018, a study published in Science reported the use of metastatic gastrointestinal cancer organoids for drug sensitivity testing [25]. This study compared and analyzed the differences in sensitivity to a series of targeted and chemotherapeutic drugs between 21 clinical patients and their corresponding PDOs, demonstrating strong consistency between the two. Compared with the patients' actual therapeutic outcomes, the PDO predictions were robust (sensitivity 100%, specificity 93%, positive predictive value 88%, and negative predictive value 100%). In 2020, Yao Y et al. [26] utilized biopsy tissues from 112 patients with locally advanced rectal cancer to construct 96 rectal cancer organoids. Eighty of these were selected to test their response to chemoradiotherapy, and the results showed that the sensitivity of rectal cancer organoids to chemoradiotherapy was highly consistent with the patients' clinical responses (sensitivity 78%, specificity 92%, accuracy 84%). Subsequently, consistency between PDO drug response and patient clinical response has also been observed in gastric cancer, breast cancer, and other tumors. Yan HHN et al. [27] established a gastric cancer organoid biobank using tumor tissues, adjacent normal tissues, and lymph node metastasis samples from 34 gastric cancer patients. Among them, two cases developed metastasis and received postoperative combination therapy with cisplatin and 5-FU, both showing good responses. Another case received preoperative chemotherapy and showed no response to postoperative capecitabine. Investigating the sensitivity of the PDOs from these three cases to the corresponding compounds revealed that the drug sensitivity of the PDOs was completely consistent with the clinical responses of the respective patients. Guillen KP et al. [28] generated PDX and PDO models from tumor samples of breast cancer patients with endocrine therapy resistance, recurrence, and metastasis, and performed histomorphological, genomic, and drug sensitivity analyses on these samples. The results indicated that both breast cancer PDX and PDO models highly recapitulated the tissue biology and genomics of their source tumors, and their responses to anti-tumor drugs were consistent. In this study, a patient with stage IIA triple-negative breast cancer developed liver metastasis approximately one year after undergoing preoperative chemotherapy and surgery. The researchers conducted in vitro and in vivo drug sensitivity tests on the constructed PDO and PDX models and found that the microtubule inhibitor eribulin had the best therapeutic effect. Based on this finding, the patient was guided to receive eribulin treatment, resulting in complete remission of the liver metastasis lasting nearly 5 months. These studies provide preliminary evidence for the potential of PDOs to guide clinical drug use for cancer patients. Additional research has shown that by comparing the drug response differences between normal organoids and PDOs, highly selective drugs can be identified, which may help reduce toxic side effects in clinical patients. Thus, conducting drug sensitivity testing via PDOs to discover the most suitable drug treatment plan will help improve clinical efficacy for cancer patients, reduce toxic side effects, the risk of drug resistance, and the likelihood of tumor progression, maximizing patient benefit.

   Therefore, leveraging patient-derived bladder cancer organoid models to conduct anti-HER2 antibody-drug conjugate sensitivity testing for locally advanced or metastatic bladder cancer, establishing a standardized bladder cancer organoid drug sensitivity testing system, and formulating screening criteria for bladder cancer organoid drug sensitivity testing, will enable the assessment of the clinical efficacy of anti-HER2 ADC therapy in these patients. This approach can assist in developing novel individualized treatment plans for clinical application and undergo multi-center clinical validation, ultimately achieving true "avatar drug testing."
2. Research Question and Objectives (Scientific Questions and Research Goals)

Research Question: This study employs a clinical controlled trial design to compare the one-year, two-year, and three-year overall survival rates between a patient group receiving interventions guided by organoid drug sensitivity testing and a patient group where treatment selection is based on HER2 protein expression levels determined by IHC. Univariate Kaplan-Meier survival analysis will be used to compare the differences in overall survival between the two groups. The study aims to evaluate the application value of tumor organoid drug sensitivity experiments in guiding anti-HER2 ADC therapy for bladder cancer.

Research Objective: By observing the clinical efficacy of anti-HER2 ADC therapy guided by the tumor organoid drug sensitivity method in bladder cancer patients, this study aims to evaluate the application value of tumor organoid drug sensitivity experiments in guiding individualized treatment with anti-HER2 ADC drugs for bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-80 years, any gender; 2. All bladder cancer patients to be included in the study must meet the inclusion criteria in item 3 regarding staging, and tumor biopsy tissue taken before ADC treatment will be used for organoid culture; 3. Patients with unresectable locally advanced (cT4b and/or N2-3) or metastatic bladder cancer (M1) who have failed platinum-based chemotherapy; 4. Patients who have shown disease progression after at least one round of platinum-based chemotherapy, or have no satisfactory alternative treatment options; 5. Patients who can tolerate adverse reactions from ADC drug enfortumab vedotin treatment; 6. ECOG performance status score of 0-2; 7. Judged by the investigator to be able to comply with the trial protocol, have good adherence, cooperate in monitoring adverse events and efficacy, and participate in follow-up; 8. Voluntarily participate in this clinical trial, understand the study procedures, and have signed the informed consent form for participation.

Exclusion Criteria:

* 1. Patients with locally advanced or metastatic bladder cancer who have not previously received platinum-containing chemotherapy; 2. Individuals with immunodeficiency or impairment (e.g., patients with AIDS, or those using immunosuppressants or undergoing radiotherapy); 3. Participants known to be allergic to the investigational drug, similar drugs, or excipients, or those with allergic constitution; 4. Individuals on long-term steroid medication or with a history of drug abuse or dependence; 5. Those who are planning to become pregnant, are currently pregnant, or are breastfeeding; 6. Individuals with abnormal blood routine, liver and kidney function, or coagulation indicators (considered abnormal if one or more of the following are met):

  1. Absolute neutrophil count (ANC) ≤ 1.5 × 10⁹/L;
  2. White blood cell count (WBC) ≤ 3.0 × 10⁹/L;
  3. Platelet count (PLT) ≤ 90 × 10⁹/L;
  4. Hemoglobin (HB) ≤ 90 g/L;
  5. Total bilirubin (TBIL) ≥ 1.5 × the upper limit of normal (ULN) of the institution;
  6. Estimated glomerular filtration rate (eGFR) ≤ 30 ml/min/1.73m²;
  7. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≥ ULN (except for patients receiving anticoagulant therapy, if considered clinically acceptable by the investigator); 7. Participants with other factors that may cause the study to be prematurely terminated, including:

  <!-- -->

  1. History or current diagnosis of myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML);
  2. History of clear neurological or psychiatric disorders, including epilepsy or dementia;
  3. Severe comorbidities that endanger patient safety or affect study completion (e.g., severe hypertension, diabetes, thyroid disorders);
  4. Other serious diseases requiring concomitant treatment, with severe laboratory abnormalities;
  5. Other serious diseases accompanied by family or social factors that could impact participant safety, or the collection of data and samples;
  6. Uncontrolled comorbid conditions, including but not limited to persistent or active infections requiring treatment, symptomatic congestive heart failure, unstable angina, or arrhythmias; 8. Participants deemed unsuitable for this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable locally advanced (cT4b and/or N2-3) or metastatic bladder cancer (M1) who have failed platinum-based chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year OS , Two-year OS and Three-year OS | 2026.01.01-2028.12.31
  One-year overall survival rate, two-year overall survival rate, three-year overall survival rate

SECONDARY OUTCOMES:
One-year PFS ,Two-year PFS and Three-year PFS | 2026.01.01-2028.12.31
  One-year progression-free survival rate, two-year progression-free survival rate, three-year progression-free survival rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes